CLINICAL TRIAL: NCT06312943
Title: "Translating Articular Biomarkers Into Diagnoses"
Acronym: ARTBioSes
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP180414; 2022-A02170-43 (Other: France : Ministry of Health)
Record Dates: First submitted 2024-01-08; First posted 2024-03-15 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Inflammatory and Non-inflammatory Bone and Joint Diseases
Keywords: Osteoarthritis; Rheumatoid arthritis; Inflammatory joint disorders; RAMAN spectroscopy; Biomarkers
MeSH Terms: conditions — Joint Diseases; Osteoarthritis; Arthritis, Rheumatoid | interventions — Histocompatibility Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Joint fluid or tissue sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with various bone and joint diseases: Patients with various bone and joint diseases
  Interventions: Other: Collection of joint fluid or tissue sample

INTERVENTIONS:
Other: Collection of joint fluid or tissue sample — During a puncture or joint surgery planned as part of the routine care of the patient, a part of the joint fluid or tissue sample will be collected in order to carry out the analyzes planned for the research.

SUMMARY:
Early diagnosis is a key factor in the prevention and management of rheumatic diseases. Rheumatic diseases are classically diagnosed based on criteria combining clinical, biological and radiological features. However, in up to 20% of the cases, diagnoses remain unstated and underlying rheumatic diseases unclassified, which might lead to delayed specific treatment and unfavourable clinical outcomes. In addition, conventional methods could lack sensitivity and specificity for early diagnosis. Biological samples are attractive targets for the early detection of articular damage because they allow for collection of multiple levels of information from the clinic and the laboratory]. Biological samples most frequently collected from patients with rheumatic diseases are synovial fluid by joint aspiration, blood by venous puncture and tissue specimen by surgery. The investigators hypothesize that in challenging situations, novel biomarkers detected from synovial fluid or articular tissues using both conventional (e.g. histology, immunodetection, PCR) and innovative (e.g. Raman spectroscopy, nanospectroscopy) laboratory tests may help refining diagnosis and better classifying patients with rheumatic diseases.

DETAILED DESCRIPTION:
Early diagnosis is a key factor in the prevention and management of rheumatic diseases. Rheumatic diseases are classically diagnosed based on criteria combining clinical, biological and radiological features. However, in up to 20% of the cases, diagnoses remain unstated and underlying rheumatic diseases unclassified, which might lead to delayed specific treatment and unfavourable clinical outcomes. In addition, conventional methods could lack sensitivity and specificity for early diagnosis. Biological samples are attractive targets for the early detection of articular damage because they allow for collection of multiple levels of information from the clinic and the laboratory. Biological samples most frequently collected from patients with rheumatic diseases are synovial fluid by joint aspiration, blood by venous puncture and tissue specimen by surgery. The investigators hypothesize that in challenging situations, novel biomarkers detected from synovial fluid, blood or articular tissues using both conventional (e.g. histology, immunodetection, PCR) and innovative (e.g. Raman spectroscopy, nanospectroscopy) laboratory tests may help refining diagnosis and better classifying patients with rheumatic diseases.

Synovial fluid is primarily composed of water, proteins, proteoglycans, glycosaminoglycans, lipids, small inorganic salts, and metabolites such as amino acids or sugars. Individual synovial fluid components may often perform multiple functions. For example, hyaluronic acid maintains the complex viscoelastic properties of synovial fluids and regulates the biological activity of advanced glycation end-products, cytokines, and enzymes associated with osteoarthritis. Normal joint function is dependent on the status of synovial fluid composition, especially considering the large interaction between the individual components. Although conventional laboratory tests have been used by rheumatologists for the past 50 years, they provide limited quantitative data and cannot specifically describe the biochemical and chemical changes, such as alterations in protein composition and proteomic profile undergone by synovial fluids in arthritic joints. Measurements that reflect the entire synovial fluid chemical, biological or viscoelastic profile could be interesting additional tools. An example of innovative measurement technique is Raman spectroscopy that can be used to detect changes in synovial fluid from patients with rheumatic diseases. Raman band intensity ratios vary significantly in spectra collected from synovial fluid in patients with radiological evidence of osteoarthritis damage. Changes to the protein secondary structure could be used as general marker of chemical changes in synovial fluid and that these changes can be associated with radiographic scoring of knee damage. Other publications focused on the Raman analysis of crystals extracted from synovial fluids. Our group developped Surface Enhanced Raman Spectroscopy (SERS) using nanoparticles that might be more sensitive than conventional Raman spectroscopy in characterizing biofluids especially the entire synovial fluid and deciphering specific rheumatic disease spectral signatures.

Blood biomarkers have long been used for the diagnosis and follow-up of rheumatic diseases. They are mainly markers of auto-immunity, inflammation, cartilage degradation or bone remodelling.

Articular tissues include articular cartilage, bone, meniscus, synovial membrane, fat, tendons, ligaments, muscles. They are obtained during surgery. Their analysis is precious to characterize auto-immunity, inflammation, cartilage degradation or bone remodelling local status and to study local activation of cellular and molecular pathways of interest using conventional techniques of cellular and molecular biology.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Inflammatory and non-inflammatory bone and joint diseases requiring synovial fluid aspiration and/or joint replacement
* Collection of non-opposition
* Affiliated to or beneficiary of social security

Exclusion Criteria:

* Inability to speak and/or read French
* Neoadjuvant therapy
* Patients under tutor or curatorship
* Protected adults,
* Patients benefiting of State Medical Aid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ¨Patients with various bone and joint diseases
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2028-10 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Tissues and biofluid spectra using surface-enhanced Raman spectroscopy | Inclusion
  Molecular signature of articular samples
Protein expression using immunodetection techniques and RNA expression using PCR | Inclusion
  Cellular signature of articular samples

SECONDARY OUTCOMES:
Tissues and biofluid spectra using surface-enhanced Raman spectroscopy | Inclusion
Protein expression using immunodetection techniques and RNA expression using PCR | Inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Christelle Nguyen, MD, PhD, Principal Investigator — Service de Médecine Physique et de Réadaptation, Hôpital Cochin
Locations (1):
- Service de Médecine Physique et de Réadaptation, Hôpital Cochin, Paris, IDF, France

IPD SHARING:
Plan to Share IPD: No